CLINICAL TRIAL: NCT02639312
Title: Natural History of Craniofacial Anomalies and Developmental Growth Variants
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160040; 16-D-0040
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: Prognathism; Retrognathism; Dentofacial Deformities
Keywords: Craniofacial; Microsomia; Mandibular; Facial Defects; Hasburg Jaw; Natural History
MeSH Terms: conditions — Prognathism; Retrognathia; Dentofacial Deformities; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: hemifacial microsomia
- 2: mandibular prognathism

SUMMARY:
Background:

Some head and facial abnormalities are rare and present at birth. Others are more common, and may not show up until puberty. These conditions have different causes and characteristics. Researchers want to learn more about these conditions by comparing people with face, head, and neck abnormalities to family members and to healthy volunteers without such conditions.

Objectives:

To learn more about abnormal development of the face, head, and neck. To determine their genetic variants.

Eligibility:

People who have not had surgery for facial trauma:

People ages 2 and older with craniofacial abnormalities (may participate offsite)

Unaffected relatives ages 2 and older

Healthy volunteers ages 6 and older

Design:

Participants will be screened with medical history and physical exam focusing on head, face, and neck

Participants may be followed for several years. Visits may require staying near the clinic for a few days.

A visit is required for the following developmental stages, along with follow-up visits:

Age 2-6

Age 6-10

Age 11-17

Age 18 and older

Visits may include:

Medical history

Physical exam

Questionnaires

Oral exam

Blood and urine tests

Cheek swab: a cotton swab will be wiped across the inside of the cheek several times.

Cone beam CT scan (CBCT): x-rays create an image of the head, face, teeth, and neck. Participants will

stand still or sit on a chair for about 20 minutes while the scanner rotates around the head.

Photos of the head and face

Offsite participants will provide:

Copies of medical and dental records

Leftover tissue samples from previous surgery

Blood sample or cheek swab

DETAILED DESCRIPTION:
Study Description:

This is a natural history study that will examine craniofacial anomalies that affect the normal development of the facial skeleton, including birth defects and dentofacial developmental abnormalities that express themselves with the growth of the individual. Craniofacial anomalies may be rare and present at birth, such as hemifacial microsomia (1 in every 7500 live births), or common, such as dentofacial deformities including the Habsburg Jaw or mandibular prognathism (1% of the US population) that becomes apparent as a child enters puberty. These are striking disorders as they involve the face and surrounding structures, which is a focal point of self-identity and are intimately tied to quality of life and daily function.

Objectives:

Primary Objective:

To characterize and determine genetic variants of rare and common craniofacial anomalies

Secondary Objectives:

1. To establish a curated craniofacial phenomic/genomic database
2. To collect data related to clinically indicated procedures and care performed at the NIH

Endpoints:

Primary Endpoint:

Phenotypic and genomic characterization of craniofacial anomalies will be performed. Phenotypes from affected subjects and healthy volunteers will be assessed using extensive clinical evaluations, 3D cone-beam computed tomography-based geometric morphometric, cephalometric analyses, and surface morphology. Genetic variants will be identified through genomic analysis and compared with genetic patterns obtained from healthy volunteers.

Secondary Endpoints:

1. To create a database with phenotypic and genetic data, collected from the long-term follow up of subjects (females and males) with craniofacial disorders and healthy volunteers
2. To link the data with their clinical information to understand the craniofacial disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

For Subjects:

* Age > 2 to < 100 with craniofacial anomalies/abnormalities. Affected family member (defined as an individual with a demonstrable relationship, any family relationship no matter how distant, with the above subject in the pedigree) who expresses craniofacial anomalies will be classified as a subject.
* Able to provide consent, or in the case of minors, have a legally authorized representative to provide consent.

For Unaffected Family Members:

* These family members are defined as individuals with a demonstrable relationship (any family relationship, no matter how distant) with a proband subject by pedigree who do not express craniofacial anomalies.
* >= 2 years old to <= 100 years old.
* Able to provide consent, or in the case of minors, have a legally authorized representative to provide consent.

For Healthy Volunteers:

* In good general health.

  ->= 6 years old to < 100 years old.
* Able to provide consent, or in the case of minors, have a legally authorized representative to provide consent.
* Absence of a craniofacial congenital anomaly or malocclusion.
* No family history of a craniofacial syndrome.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

For All Participants:

* A history of facial trauma requiring surgical treatment and facial reconstruction.
* Refusal for both genetic testing and CBCT imaging. Participants must agree to at least one of the two (one or the other is required to participate).

For Healthy Volunteers:

-Female volunteers who are pregnant or nursing.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: -Subjects w/craniofacial anomalies or dentofacial deformities -Families of subjects with craniofacial anomalies or dentofacial deformities -Case Controls
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2046-12-31 (Estimated); Study Completion 2046-12-31 (Estimated)

PRIMARY OUTCOMES:
Database or registry | 17 years
  using both extensive clinical evaluations, 3D cone-beam computed tomography-based geometric morphometric and cephalometric analyses, and surface morphology

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinia Almpani, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Proffit WR, Fields HW Jr, Moray LJ. Prevalence of malocclusion and orthodontic treatment need in the United States: estimates from the NHANES III survey. Int J Adult Orthodon Orthognath Surg. 1998;13(2):97-106. PMID 9743642
- [Background] Cruz RM, Krieger H, Ferreira R, Mah J, Hartsfield J Jr, Oliveira S. Major gene and multifactorial inheritance of mandibular prognathism. Am J Med Genet A. 2008 Jan 1;146A(1):71-7. doi: 10.1002/ajmg.a.32062. PMID 18074368
- [Background] Frazier-Bowers S, Rincon-Rodriguez R, Zhou J, Alexander K, Lange E. Evidence of linkage in a Hispanic cohort with a Class III dentofacial phenotype. J Dent Res. 2009 Jan;88(1):56-60. doi: 10.1177/0022034508327817. PMID 19131318
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-D-0040.html